CLINICAL TRIAL: NCT00417261
Title: A Randomized, Double-Blind, Placebo-Controlled, Active Comparator, Ascending Single and Multiple Dose, Seamless Design Study to Explore the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Two Orally Administered Compounds, ATF936 and AXT914, in Healthy Male and Female Subjects
Brief Title: Safety, Tolerability, Pharmacodynamic and Pharmacokinetic Effects of Single and Multiple-Doses of ATF936 and AXT914 Administered Orally in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CATF936A2201
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: ATF936, AXT914, healthy subjects, pharmacokinetics, parathyroid hormone, osteoporosis; Healthy male and female subjects
MeSH Terms: conditions — Osteoporosis | interventions — ATF936; AXT914

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): ATF936
  Interventions: Drug: ATF936
- 2 (Experimental): AXT914
  Interventions: Drug: AXT914
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: ATF936; Drug: AXT914

INTERVENTIONS:
Drug: ATF936
  Arms: 1; 3
Drug: AXT914
  Arms: 2; 3

SUMMARY:
This is a first-in-human study and is designed to evaluate the safety, tolerability, pharmacodynamic and pharmacokinetic effects of a single and multiple-doses of ATF936 and AXT914 administered orally in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Study population:

Open-label safety cohort, Phases A and B: Healthy male and female subjects between the ages 18 to 68 years (inclusive), in good health as determined by past medical history, physical examination, vital signs assessments, electrocardiograms, routine laboratory testing (hematology, biochemistry, urinalysis) and the opinion of the investigator at screening and baseline. Female subjects must be of non-childbearing potential who are either surgically sterilized or are post-menopausal (see inclusion criterion #2 below)

Phase C: Healthy post-menopausal females of up to and including 68 years of age, in good health as determined by past medical history, physical examination, vital signs assessments, electrocardiograms, routine laboratory testing (hematology, biochemistry, urinalysis) and the opinion of the investigator at screening and baseline.

All Phases:

* Post menopausal status is established according to the following guidelines:

  * Cessation of menses for ≥ 3 years.
  * Documented total hysterectomy/bilateral oophorectomy at least 2 years prior to study participation.
  * Cessation of menses for < 25 years.
  * FSH level > 30 IU/L (confirmed prior to dosing).
  * All female subjects, regardless of age, must have negative pregnancy test results at screening and at each baseline.
* At screening and initial baseline, Vital signs in supine position should be within the following ranges: Oral body temperature: 35.0-37.5 °C (inclusive), Systolic blood pressure: 80 - 150 mm Hg (inclusive), Diastolic blood pressure: 50 - 90 mm Hg (inclusive), Pulse rate: 40 - 90 bpm (inclusive)
* Subjects must weigh at least 60 kg to participate in the study.
* Body Mass Index:

  * Open-label safety cohort, Phases A and B: Subjects must have a body mass index (BMI) within the range of 18 to 28 kg/m2, inclusive (a BMI of up to 30 kg/m2 is permissible only if it can be demonstrated that recruitment is being hindered by having an upper limit of 28 kg/m2).
  * Phase C: Subjects must have a body mass index (BMI) strictly within the range of 18 to 28 kg/m2 (inclusive).
* Vitamin D 25-(OH) serum level of ≥ 15 ng/ml (for subjects in Phase C at Screening only).

All Phases:

* Normocalcemia - serum calcium ≥ 8.5 mg/dL and ≤ 10.2 mg/dL (or according to local lab ranges).

Exclusion Criteria:

All phases:

* Smokers (use of tobacco products in the previous 3 months). Smokers will be defined who reports tobacco use and/or who has a urine cotinine ≥ 300 ng/ml.

Open-label safety cohort, Phases A and B:

* Use of prescription and non-prescription medications:

Open-label safety cohort, Phases A and B: Use of any prescription drugs within 4 weeks prior to study start, and/or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements included) within 2 weeks prior to study start. If needed, acetaminophen is acceptable.

Phase C: Use of any prescription and/or non-prescription drugs (including vitamins, herbal supplements, and dietary supplements) within 4 weeks prior to study start, unless otherwise specified. If needed, acetaminophen is acceptable.

* Subjects who are using or have used within the last 2 months, any medicine in one or more of the following classes (Phase C only): An HMG coA reductase inhibitor ("statin"), a thiazide-type diuretic, an alpha adrenergic blocker, an anticonvulsant (for example, diphenylhydantoin, phenobarbital or carbamazepine) or a heparin class anticoagulant.

All Phases (pertaining primarily to post-menopausal females):

* Subjects who are using or have used any medicine in one or more of the following classes:

  * Within the last 3 months: Estrogens, Hormone replacement therapy including Selective Estrogens Receptor Modulators (SERMs)
  * Within the last 12 months: Strontium ranelate, PTH, Calcitonin, Aluminum supplements
  * Within the last 24 months: Bisphosphonates (no bisphosphonate use permitted in last 24 months)
* Subjects with a history of chronic use of systemic corticosteroids (oral or i.v.) within the last year where the total dose exceeds 750 mg of oral prednisone or equivalent. [NOTE: Use of corticosteroids in forms such as topical creams, nasal or inhaled formulations or those injected locally (intra-articular) more than one month prior to screening are NOT exclusionary].
* Subjects with cancer or history of malignancy of any organ system, treated or untreated, at any time, whether or not there is evidence of local recurrence or metastases. [NOTE - the following exceptions will apply: Basal cell or squamous cell carcinoma of the skin or colonic polyps with non-invasive malignancy that have been removed and not recurred, and carcinoma in-situ (CIS) of either the breast, cervix or uterus that has been surgically removed and has not recurred].
* History or clinical evidence of abnormal thyroid function or thyroid disease (hypo-or-hyperthyroidism, TBG deficiency, etc.) or other endocrine disorders or conditions.
* Subjects with bony deformities and/or neuromuscular irritability indicative of chronic hypocalcaemia.
* Subjects with a history or evidence of previous/recent (within 6 months) fractures.
* Participation in any clinical investigation within 4 weeks prior to initial dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 ml or more of blood or plasma within 8 weeks prior to initial dosing, or longer if required by local regulation.
* History or clinical evidence of any bleeding disorders (i.e., poor coagulation, prolonged clotting time, etc.) at Screening and/or initial Baseline.
* Hemoglobin of < 12 g/dL at Screening and/or initial Baseline.
* Significant illness within 2 weeks prior to initial dosing.
* A past medical history of clinically significant ECG abnormalities or a family history (grandparents, parents and siblings) of prolonged QT-interval syndrome.
* Any Surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study, including bowel, gastrointestinal, renal, pulmonary, pancreatic, hepatic, hematological, immunological, or neurological disorder.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2006-11; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Phase A: Safety and tolerability of single, oral doses of ATF936 and AXT914 under proposed conditions in healthy male and female subjects. Pharmacokinetics (PK) and pharmacodynamics (PD) of ATF936 and AXT914 in healthy male and female subjects.
Phase B: A head-to-head comparison of ATF936 and AXT914, each given at its pharmacologically effective dose as determined in Phase A.
Phase C: Similarity of PK/PD profile to single-dose profile after limited multiple dosing in healthy post-menopausal females. Early bone biomarker information after multiple dosing for best candidate as selected in Phase A or Phase B

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States